CLINICAL TRIAL: NCT03049228
Title: Cardiac Mitochondrial Function: Comparison of in and ex Vivo Measurements
Brief Title: In and ex Vivo Mitochondrial Function of the Heart
Acronym: 31P
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Diabetes Fonds (Other)
Responsible Party: Sponsor
Other Study IDs: NL.ABR.48376
Record Dates: First submitted 2017-01-25; First posted 2017-02-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies
Keywords: Spectrum Analysis; Mitochondria; Peroxisome Proliferator-Activated Receptors; Respirometry; Human; Heart
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies | interventions — Hematologic Tests; Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — From a fasting blood sample will DNA be extracted from leucocytes to study genetic variants that may affect results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 Diabetic Patients: * Obese (BMI > 27 kg/m2 < 35 kg/m2)
  * Non-insulin dependent; they must be on sulphonylurea(SU)- derivate or metformin therapy for at least six months with a constant dose for at least two months, or on dietary treatment for at least six months
  * They should have a (moderately) well-controlled diabetes (defined by a HbA1c<8%)
  Interventions: Diagnostic Test: 31P-MRS scan and cardiac MRI scan; Diagnostic Test: Atrial biopsy for high-resolution respirometry; Diagnostic Test: Blood analysis; Diagnostic Test: Body composition; Diagnostic Test: Indirect Calorimetry
- Obese Subjects: * A similar BMI as T2DM patients (BMI > 27 kg/m2< 35)
  * Normo-glycemic with fasting plasma glucose levels lower than 6,1 mmol/L.
  Interventions: Diagnostic Test: 31P-MRS scan and cardiac MRI scan; Diagnostic Test: Atrial biopsy for high-resolution respirometry; Diagnostic Test: Blood analysis; Diagnostic Test: Body composition; Diagnostic Test: Indirect Calorimetry
- Lean subjects: * BMI between 20-25 kg/m2
  * Normo-glycemic with fasting plasma glucose levels lower than 6,1 mmol/L.
  Interventions: Diagnostic Test: 31P-MRS scan and cardiac MRI scan; Diagnostic Test: Atrial biopsy for high-resolution respirometry; Diagnostic Test: Blood analysis; Diagnostic Test: Body composition; Diagnostic Test: Indirect Calorimetry

INTERVENTIONS:
Diagnostic Test: 31P-MRS scan and cardiac MRI scan — 31P-MRS measurement of the heart: Phosphorous magnetic resonance spectroscopy (31P-MRS) will be used for the determination of the energy status of the heart in vivo. The localization of phosphorus energy metabolites in the heart will be performed by one-dimensional spectroscopic imaging, resulting in spectra from slices through the heart of 1 cm thickness. The peaks of PCr and ATP will be fitted in order to calculate the ATP/PCr ratio.
  The measurement of cardiac function is a standardised protocol. In the 4 chamber view setting a T1 mapping sequence will be performed for the detection of fibrosis. Hereafter patients will receive contrast for T2 mapping and late enhancement studies for determining extracellular volume and ischemia.
  Other Names: Spectrum Analysis; MRI
Diagnostic Test: Atrial biopsy for high-resolution respirometry — Mitochondrial respiration rates are ex vivo measured in tissue homogenates under exposure of different substrates, stimulating different complexes of the electron transport chain of the mitochondria.
  Other Names: Oxygraph
Diagnostic Test: Blood analysis — To determine blood glucose metabolism and renal function.
Diagnostic Test: Body composition — This device uses air displacement plethysmography for determining percent fat and fat-free mass in adults and children. The 5-minute test consists of measuring the subject's mass (weight) using a very accurate electronic scale, and volume, which is determined by sitting inside the BOD POD chamber. From these two measurements, the subject's body composition is calculated.
  Other Names: BodPod
Diagnostic Test: Indirect Calorimetry — As basal energy metabolism might be related to cardiac metabolism and mitochondrial function, and basal metabolic rate shows inter-individual variance, it is an important subject characteristic of the patients. Resting substrate oxidation rates are measured with indirect calorimetry for 30 minutes. A ventilated hood is connected to indirect calorimetry equipment, which measures concentrations of oxygen consumption and CO2 production. From these parameters, the respiratory quotient (RQ), as well as energy expenditure and substrate metabolism will be computed. During this measurement, every 10 minutes (so 4 times) one tube of blood (10ml) will be drawn for the analysis of lipid and glucose metabolites.
  Other Names: Ventilated Hood; Basal energy metabolism; Omnical

SUMMARY:
It has been suggested that mitochondrial dysfunction might play a role in the development of diabetic cardiomyopathy. From animal studies, it has been suggested that an altered PPAR and PGC1 expression is involved in the reduced cardiac mitochondrial function, however human data on cardiac mitochondrial function and PPAR regulation is scarce. The latter is due to the fact that there is no validated measurement for assessing cardiac mitochondrial function non-invasively in vivo. It has been suggested that measuring PCr/ATP ratio with 31P-MRS in the heart reflects cardiac mitochondrial function. However, so far no direct validation of this method has been performed. The aim of this study will be to validate in vivo 31P-MRS with ex vivo measurements of mitochondrial function. To this end, the hypothesis is that in vivo 31P-MRS is a valid method for measuring cardiac mitochondrial function when compared with ex vivo mitochondrial respirometry.

DETAILED DESCRIPTION:
Cardiovascular diseases remain the main cause of death in type 2 diabetes. Most of this is attributed to atherosclerosis and elevated blood pressure, though even when corrected for these factors, patients with type 2 diabetes are still at increased risk for developing cardiac failure, mainly through diastolic dysfunction. This phenomenon has also been described as diabetic cardiomyopathy. Although not much is known about the aetiology of this disease, there is compelling evidence from animal research that an increased intracellular cardiac fat accumulation and mitochondrial dysfunction, as seen in type 2 diabetes, may play a part in this development.

The reason for a reduced mitochondrial function in diabetic cardiomyopathy is not completely understood, however the gene regulatory pathway of peroxisome proliferator-activated receptor alpha (PPAR-α) has been identified as an important determinant of the shift in substrate metabolism and regulation of oxidative metabolism in type 2 diabetes. In animal studies, the role of PPARα has been tested extensively. In mice with cardiac-restricted overexpression of PPARα (MHC-PPAR), it was found that PPAR-α is involved in the upregulation of CPT-1 in mitochondria, which increases the uptake of long-chain fatty acid into mitochondria and facilitates the fatty acids to undergo beta-oxidation. Chronic exposure to elevated FFAs down regulates PPAR-α in rodent cardiomyocytes, which would further decrease cardiac function by inhibition of FA oxidation and increased intracellular fat accumulation. It is therefore speculated that the increase in fatty acid availability in type 2 diabetes and obesity (due to excessive fat mass) leads to a decrease in cardiac PPAR-α metabolism and thereby a decrease in mitochondrial metabolism, which in turn is paralleled by an increased cardiac fat accumulation and cardiac lipotoxicity.

So far, human studies on PPAR expression in the heart are scarce. Marfella et al. found unaltered expression of PPAR-α in patients with the metabolic syndrome. Conversely, Anderson et al., showed a slightly reduced PPAR-α protein level and a slightly higher PGC1α level in diabetic atrial tissue, though these differences did not reach statistical significance in this cohort of patients. As this study was performed in a small group of subjects and failed to determine the down-stream targets of the PPAR metabolism or mitochondrial function, it remains unclear whether like in animal studies also in humans a reduced PPAR-a expression is related to mitochondrial dysfunction. Therefore there is need for studies exploring the role of PPAR-a in human heart and the connections with oxidative metabolism and cardiac function. Mice lacking the cardiac lipase ATGL (ATGL-/- mice) was actually due to a reduction in PPAR metabolism, and that the cardiomyopathy in these mice could be completely prevented by treating these animals with synthetic PPAR-a ligands. Very interestingly, patients with a mutation in the same ATGL gene are also characterized by excessive cardiac and muscle fat accumulation and reduced mitochondrial function. Treating two patients with such mutations (which is a very rare mutation) with a PPAR-agonist (bezafibrate) resulted in improved mitochondrial function and a reduction in muscle and cardiac lipid accumulation. These data support the notion that a disturbed PPAR metabolism may be involved in the development of cardiomyopathy, also in humans. However, unfortunately, there is limited data on PPAR-expression in the failing human diabetic heart. Therefore there is need of studies validating these mechanisms in humans, as these findings might have great consequences; prevention and treatment of cardiac lipid accumulation with drugs that improve mitochondrial function, such as PPAR-agonists, might be of value to patients with type 2 diabetes. Also in other cardiac diseases, such as chronic heart failure and ischemic heart disease, it has been suggested that fat accumulation and mitochondrial dysfunction may play a role, which means that these patients might benefit as well from treatment with drugs that target mitochondrial function.

Although there is compelling evidence that mitochondrial function plays an important role in cardiac metabolism, measuring cardiac mitochondrial function non-invasively in vivo remains a challenge. In vivo mitochondrial function can be estimated non-invasively with 31P-Magnetic Resonance Spectroscopy (31P-MRS), whereby the ratio Phospho-creatine (PCr) over Adenosine Triphosphate (ATP) is measured (PCr/ATP-ratio). Several studies have shown that this ratio is reduced in patients with type 2 diabetes, and that a low PCr/ATP ratio predicts mortality in patients with cardiac failure15-17. In skeletal muscle it has been shown that PCr-resynthesis strongly correlates with mitochondrial oxidative capacity18. However, if this method in the heart truly reflects mitochondrial function in humans has not been revealed.

In 31P-MRS a 2 dimensional measurement method is used, in which multiple slices are planned over the heart. One slice is planned directly at the base of the heart in the plane just below the valves and contains both ventricular and septal tissue of both chambers. Here the signal for acquisition of the spectrum will be derived. This method can be validated against the golden standard for mitochondrial function: ex vivo respirometry of cardiac tissue19. Thus, mitochondrial respiration rates are measured in tissue homogenates under exposure of different substrates, stimulating different complexes of the electron transport chain of the mitochondria. One issue is that mitochondrial respiration may differ between atrial and ventricular tissue. However, despite the differences in absolute respiration rates, the behaviour of the different complexes and relative respiration rates (between complexes) has been shown to be very strongly related19. Since it is relatively easy to obtain atrial appendage cardiac tissue during surgery, the investigators propose to use atrial tissue obtained during surgery to validate 31P-MRS as a tool to determine mitochondrial function. The investigators will use a broad range of patients to guarantee a range in cardiac mitochondrial functions, and to examine if cardiac mitochondrial function is indeed reduced in type 2 diabetic patients.

However, as the 31P-MRS still is a technique in development and the distance to the receiver coil is crucial for obtaining spectra of good quality, the investigators intend to only include men at this time (as increased breast mass in women may decrease signal to noise ratios and hence spectral quality for analysis). Therefore, the validation of this method will only apply for the male population in this study.

ELIGIBILITY:
Inclusion Criteria:

* All patients that undergo either valve replacement surgery or a cardiopulmonary bypass procedure can be included in this study.

General inclusion criteria:

* aged between 40-75 years
* stable dietary habits (no weight loss/gain >5kg in the last 3 months)
* stable physical activity levels for at least 6 months

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* Insulin dependent T2DM subjects can not be included.
* Patients with instable angina or heamodynamically instable patients cannot be included in the study.
* Patients that use Thiazolidines (glitazone/rosiglitazone/pioglitazone/troglitazone) can not be included.
* Patients with weight gain/loss > 5 kg in the last 3 months can not be included.
* Patients with signs of cachexia (Body mass index (BMI) < 20 kg/m2 or substantial weight loss (>5%) in last 6-12 months (weight loss should be mainly non-oedematous))
* Patients with poor renal function (defined as a MDRD < 60) can not be included in the cardiac late enhancement measurements (as they can not receive contrast), though they will be included in the study for all other measurements.
* Participants with contraindications for MRI scans:

  * Electronic implants such as pacemakers or neurostimulator
  * Iron-containing corpora aliena in eyes or brain
  * Some hearing aids and artificial (heart) valves which are contraindicated for MRS
  * Claustrophobia
* Subjects, who do not want to be informed about unexpected medical findings, or do not wish that their physician is informed, cannot participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As patients will have to undergo surgery to obtain cardiac tissue for these ex vivo measurements, the investigators will only use patients that are scheduled for cardiac surgery (either for valve replacement or a cardiopulmonary bypass procedure).
  Obese type 2 diabetic patients will be compared with obese and lean normo-glycemic patients. As all patients will undergo the same measurements, this study is designed as an observational case-control study. The investigators have chosen to include both obese and lean participants, as the investigators expect that bodyweight and intra-cellular lipid accumulation affects cardiac mitochondrial function. This will probably result in a large range in mitochondrial function, which facilitates the validation of the methods.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Cardiac energy status in vivo | 1 week before surgery the patient will undergo the MRS scan. That same week the investigators will analyse the ATP/PCr ratio. Data will be presented through study completion, an average of 2 years.
  Measured with 31P-MRS to determine ATP/PCr ratio and ex vivo mitochondrial function measured with high-resolution respirometry as a golden standard to validate the in vivo MRS.
Cellular respiration ex vivo | At surgery the investigators obtain tissue samples. Within an hour the investigatorswill use the oxygraph to measure the cellular respiration. Data will be presented through study completion, an average of 2 years.
  With the oxygraph the investigators measure how well the muscle is capable of oxidative phosphorylation which reflect the mitochondrial function. This reflects the mitochondrial capacity.

SECONDARY OUTCOMES:
Cardiac function | 1 week before surgery the patient will undergo the MRI scan. The investigators will analyse this scan within a week. Data will be presented through study completion, an average of 2 years.
  With MRI the investigators will determine systolic (ejection fraction) and diastolic function.
Cardiac lipid accumulation | 1 week before surgery the patient will undergo the MRS scan. The investigators will analyse this scan within a week. Data will be presented through study completion, an average of 2 years.
  The investigators will measure cardiac lipid accumulation ex vivo from tissue (Elektron Microscopy) and in vivo with MRI.
Role of PPAR metabolism in the heart on the development of diabetic cardiomyopathy | The investigators will obtain tissue samples from surgery. The investigators will analyse this tissue within a week. Data will be presented through study completion, an average of 2 years.
  With the use of the tissue the investigators will determine cardiac PPAR expression and possible down-stream targets involved in mitochondrial metabolism ex vivo
Glucose Metabolism Status | At inclusion the investigators will take some serum and analyse it the same day. The inclusion will be around 1 week before MRI-scan and 2 weeks before surgery. Data will be presented through study completion, an average of 2 years.
  At screening the investigators will take blood samples to determine fasting blood glucose so the investigators can divide the participants between normo-glycemic and diabetes.
Height in meters | At inclusion the investigators will determine their height, this will be around 1 week before MRI-scan and 2 weeks before surgery. Data will be presented through study completion, an average of 2 years.
  To be able to determine their BMI (kg/m^2) the investigators have to measure the participants' height in meters at screening.
Weight in kilograms | At inclusion the investigators will determine their weight, this will be around 1 week before MRI-scan and 2 weeks before surgery. Data will be presented through study completion, an average of 2 years.
  To be able to determine their BMI (kg/m^2) the investigators have to measure the participants' weight in kilograms at screening.
Body composition | The investigators will measure the body composition right before the MRI-scan, this will be around 1 week before surgery. Data will be presented through study completion, an average of 2 years.
  With the Bodpod the investigators will measure the body composition of the participant.
Basal energy metabolism | The investigators will measure the basal energy metabolism right before the MRI-scan, this will be 1 week before surgery. Data will be presented through study completion, an average of 2 years.
  With the Omnical (Ventilated Hood) the investigators will measure the basal energy metabolism status of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Prof., Principal Investigator — Maastricht University
Locations (1):
- Human Biology, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided